CLINICAL TRIAL: NCT00448682
Title: A Phase II Study of Weekly 24-hour Infusion 5-fluoro-deoxyuridine (FUdR)/Leucovorin With Oxaliplatin and Docetaxel (Taxotere) as First-line Treatment in Patients With Metastatic Gastric Adenocarcinoma (IIT# 14065)
Brief Title: Combination Chemotherapy as First-Line Therapy in Treating Patients With Stage IV Gastric Cancer That Cannot Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040005; SCCC-2003150 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20050983 (Other: Western Insitutional Review Board)
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Gastric Cancer
Keywords: recurrent gastric cancer; stage IV gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Floxuridine; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FUdR + Leucovorin + Oxaliplatin + Docetaxel (Taxotere) (Experimental): Treatment will be administered on an outpatient basis. Chemotherapy will be administered weekly, 3 out of 4 weeks, on days 1, 8 and 15:
  Day 1 and Day 15 Chemotherapy Administration: Patients will be administered oxaliplatin (85 mg/m2) and docetaxel (25 mg/m2) followed by FUdR/Leucovorin (110 mg/kg//500 mg/m2) on Day 1 and Day 15 of each cycle.
  Day 8 Chemotherapy Administration On Day 8, treatment will consist of docetaxel (25 mg/m2) followed by FUdR/Leucovorin (110mg/kg//500mg/m2).
  There will be no treatment delivered week 4 (Day 22). For the purpose of this study, one cycle equals four weeks. There will be a maximum of 6 cycles.
  Interventions: Drug: Docetaxel; Drug: Floxuridine; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Docetaxel
  Other Names: Taxotere
Drug: Floxuridine
  Other Names: 5-fluorodeoxyuridine; 5-FU; FudR
Drug: Leucovorin
  Other Names: Folinic acid; Leucovorin calcium
Drug: Oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as floxuridine, leucovorin, oxaliplatin, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works as first-line therapy in treating patients with stage IV gastric cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate in patients with unresectable stage IV gastric adenocarcinoma treated with floxuridine, leucovorin calcium, oxaliplatin, and docetaxel as first-line treatment.

Secondary

* Determine the feasibility of this regimen in managing patients with unresectable stage IV gastric adenocarcinoma who have not received prior chemotherapy for metastatic disease.
* Determine disease-free survival of patients treated with this regimen.
* Evaluate overall survival of patients treated with this regimen.
* Assess the safety and toxicity of this regimen in these patients.

OUTLINE: Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and docetaxel IV over 30 minutes, floxuridine IV over 24 hours, and leucovorin calcium IV over 24 hours on days 1, 8, and 15. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 26 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed gastric adenocarcinoma meeting the following criteria:

  * Stage IV disease OR stage III disease that was re-staged as metastatic disease at time of surgery
  * Unresectable disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* Creatinine ≤ 1.5 mg/dL
* Alkaline phosphatase (AP), AST, and ALT must meet 1 of the following criteria:

  * AP normal AND AST and ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST and ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST and ALT normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No peripheral neuropathy > grade 1
* No history of severe hypersensitivity reaction to platinum agents (e.g., cisplatin or carboplatin), fluoropyrimidines, or drugs formulated with polysorbate 80
* No concurrent serious illness that would preclude study treatment or compliance
* No active infections requiring intravenous antibiotic therapy
* No other malignancy within the past 5 years except for cervical carcinoma in situ, breast ductal carcinoma in situ, colonic polyp, or squamous cell or basal cell carcinoma of the skin
* No clinically significant uncontrolled cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease, or cardiac arrhythmias) or myocardial infarction within the past 12 months

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy for metastatic gastric carcinoma
* No prior chemotherapy for metastatic gastric carcinoma

  * Prior neoadjuvant or adjuvant chemotherapy and/or radiotherapy allowed if completed therapy at least 12 months before study enrollment

    * Chemotherapy may have included taxane, platinum, or fluoropyrimidine-based regimen
* At least 2 months since prior surgery and recovered
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bach Ardalan, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FUdR + Leucovorin + Oxaliplatin + Docetaxel: Treatment will be administered on an outpatient basis. Chemotherapy will be administered weekly, 3 out of 4 weeks, on days 1, 8 and 15:
  Day 1 and Day 15 Chemotherapy Administration: Patients will be administered oxaliplatin (85 mg/m2) and docetaxel (25 mg/m2) followed by FUdR/Leucovorin (110 mg/kg//500 mg/m2) on Day 1 and Day 15 of each cycle.
  Day 8 Chemotherapy Administration On Day 8, treatment will consist of docetaxel (25 mg/m2) followed by FUdR/Leucovorin (110mg/kg//500mg/m2).
  There will be no treatment delivered week 4 (Day 22). For the purpose of this study, one cycle equals four weeks. There will be a maximum of 6 cycles.
Period: Overall Study
Arm/Group | FUdR + Leucovorin + Oxaliplatin + Docetaxel
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FUdR + Leucovorin + Oxaliplatin + Docetaxel
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 62 [39 to 85]
Gender [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Clinical Response
Description: Number of patients achieving complete response (CR) or partial response (PR) according to RECIST Criteria version 1.0.
Time Frame: 1 year
Population: The study data has not been analyzed.
Arm/Group | FUdR + Leucovorin + Oxaliplatin + Docetaxel
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Rate of Survival
Description: Patients will be followed for overall survival from date of enrollment to date of death or last contact. The extent of follow up will be described by the range and median for deceased patients and for those alive at last follow up. We will estimate the 1 year survival rates by the Kaplan-Meier method.
Time Frame: 1 year
Population: The study data has not been analyzed.
Arm/Group | FUdR + Leucovorin + Oxaliplatin + Docetaxel
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing adverse events within 1 year of receiving combination therapy of FUDR + Leucovorin + Oxaliplatin + Docetaxel for metastatic gastric adenocarcinoma.
Time Frame: 1 year
Population: The study data has not been analyzed.
Arm/Group | FUdR + Leucovorin + Oxaliplatin + Docetaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Serious and non-serious adverse events were not collected/assessed.
Arm/Group | FUdR + Leucovorin + Oxaliplatin + Docetaxel
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the University of Miami Institutional Review Board. The results have not been analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes